CLINICAL TRIAL: NCT03332524
Title: Phase II Multicenter, Double-blinded Clinical Trial of SP160412 in the Temporary Relief of Mild to Moderate (i.e,First Degree) Sunburn
Brief Title: Clinical Trial of the Safety and Efficacy of SP160412 in the Temporary Relief of Mild to Moderate Sunburn
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to stop for lack of efficacy
Sponsor: Sephoris Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16CMCL249
Record Dates: First submitted 2017-10-02; First posted 2017-11-06 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Sunburn
Keywords: 1st degree burn
MeSH Terms: conditions — Sunburn | interventions — Chlorpheniramine; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Multi-centers double-blinded clinical trial with one intervention arm with SP160412 (Ibuprofen and Chlorpheniramine combined) with one arm with Active control (Ibuprofen with placebo) and a third arm (Chlorpheniramine with Placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 Product SP160412 (Experimental): oral route, 9 doses (Capsule) of SP160412 (Ibuprofen 400 mg and Chlorpheniramine maleate 4 mg combined) in the 72 hours-period from first dose to last dose.
  Interventions: Drug: SP160412 Ibuprofen 400 mg and Chlorpheniramine maleate 4 mg
- capsules Ibuprofen&placebo (Placebo Comparator): 2 capsules Ibuprofen and 1 placebo, oral route, 9 doses of Ibuprofen 400 mg with Placebo (Capsule) in the 72 hours-period from first dose to last dose,
  Interventions: Drug: 2 capsules Ibuprofen and 1 placebo
- Capsule Chlorpheniramin&placebo (Placebo Comparator): capsule Chlorpheniramine 4mg and 1 Placebo, 3/72 hours-period from first dose to last dose, oral route
  Interventions: Drug: capsule Chlorpheniramine 4mg and 1 Placebo

INTERVENTIONS:
Drug: SP160412 Ibuprofen 400 mg and Chlorpheniramine maleate 4 mg — 2 Ibuprofen and capsules Chlorpheniramine maleate 3 time per day for 72 hours
  Other Names: 2 Capsules Ibuprofen and one capsules Chlorpheniramine
  Arms: Arm 1 Product SP160412
Drug: 2 capsules Ibuprofen and 1 placebo — Ibuprofen and placebo
  Other Names: Capsule with Ibuprofen 400 mg with Placebo
  Arms: capsules Ibuprofen&placebo
Drug: capsule Chlorpheniramine 4mg and 1 Placebo — Chlorpheniramine 4mg and one capsule Placebo 3/72days
  Other Names: Active comparator Chlorpheniramine 4 mg with Placebo
  Arms: Capsule Chlorpheniramin&placebo

SUMMARY:
A phase II multicenter, double-blinded clinical trial of the safety and efficacy of

SP160412 in the temporary relief of mild to moderate, (i.e. first degree) sunburn

DETAILED DESCRIPTION:
The objectives of the trial or study, its endpoints, its assumptions and its variables are described below:

Objectives and endpoints Study objectives

The study intends to determine and compare the safety and synergistic efficacy of the combined dosing of Ibuprofen and Chlorpheniramine maleate vs. each of the individual drugs in subjects with mild to moderate ( 1st degree) sunburn.

ELIGIBILITY:
Inclusion Criteria:

* enter the study, a participant must meet all the following criteria:

  1. Male or female, with a minimum age of 18 years old.
  2. Participant who has experienced sunburn in the past 18 hours before inclusion in the study.
  3. Participant who is willing and able to give written informed consent and understand the language used at the investigation site.
  4. Participant who is willing and able to administer the investigational medicinal product (IMP) as directed, comply with study instructions and commit to all the follow-up visits for the duration of the study.
  5. Participant with a Fitzpatrick skin type I, II or III as clinically defined by the investigator.
  6. Participant with a clinical assessment of sunburn score of 2 (mild) or 3 (moderate) according to clinical grading described in Appendix II.2. Clinical Assessment of Sunburn (page 78).
  7. Participant who is in good general health and free of any disease state or physical condition except sunburn that might impair the clinical evaluation of erythema, pain and pruritus associated with sunburn.
  8. Participant who confirms not having used sunscreen or any other lotion on the zone of investigation before the acquired sunburn and inclusion in the study.
  9. Participant who agrees not to expose themself further to the sun and not to apply any topical product (sunscreen, aftersun products, products containing aloe vera, moisturizing products…) on the zone of investigation within 18 hours before sunburn and during the study.
  10. If participant is a woman of childbearing potential and declares to be sexually active, she must have a negative urine pregnancy test (UPT) at inclusion and agree to use an effective form of birth control for the duration of the study (e.g., stable dose of oral contraceptives for at least three months before the start of the study, implant, injection, IUD, patch, NuvaRing, condom and spermicidal or diaphragm and spermicidal). Abstinence is an acceptable form of birth control for participants who are sexually active.

      Exclusion Criteria:

  <!-- -->

  1. Participant who routinely subjects himself/herself to natural or artificial tanning or the like which, in the investigator's opinion, exposes the participant to an unacceptable risk when taking part in the study.
  2. Participant who is pregnant or lactating, or is planning to become pregnant during the study.
  3. Participant who is currently enrolled in an investigational product or device study.
  4. Participant who has used an investigational product or investigational device treatment within 30 days prior to the start of the study.
  5. Participant with a medical condition (including previous history of cardiac disease, renal disease, gastrointestinal bleeding, uncontrolled hypertension) or a medication which, in the clinical investigator's judgement, makes the participant ineligible or places the participant at undue risk during the study.
  6. Participant who has a history of drug allergy or sensitivity to NSAIDs, including Aspirin, and/or to Chlorpheniramine maleate, and/or to any of the components of the IMP.
  7. Participant who has used pain relieving and/or analgesic medications (e.g. NSAIDs, ASA, opiates, Tramadol, arnica, products containing aloe vera) or psychoactive substances (e.g. marijuana) within 7 days before the start of the study.
  8. Participant who has used any topical or oral antihistamine/anti-allergy medications within 7 days prior to the start of the study.
  9. Participant who has used any photosensitizing medication (e.g., topical or systemic retinoids, tetracycline or derivatives, etc.) within 30 days of the start of the study. Estrogens as part of birth control agents or hormone replacement therapy are allowed.
  10. Participant with acute or chronic pain condition.
  11. Participant suffering from asthma.
  12. Participant who has a history of any light-sensitive disorder including but not limited to lupus erythematosus, polymorphous light eruption or porphyria.
  13. Participant with a personal or family history in a first-degree relative of malignant melanoma, dysplastic nevi or non-melanoma skin cancer.
  14. Participant who has received more than one sunburn in the last 6 months in the same zone as the study sunburnt evaluation zone.
  15. Participant who has received sunburn or other erythematous skin reaction to light within 21 days prior to the start of the study.
  16. Participant with extensive body hair, tattoos or other adornment that would make clinical assessments difficult.
  17. Participant who is known to be noncompliant or is unlikely to comply with the requirements of the study protocol in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Self reported pain score on Pain Numeric Scale (NRS) at each visit | Twice a day (in the morning and at night) from day 1 to day 5
  To measure the efficacy of SP160412 in the reduction of pain as reported by the participants. The Brief Pain Inventory - short version assesses pain in the last 24 hours and its impact on daily functioning. It evaluates the worst, the least, the average pain the participants felt during the last day and the actual pain. Scores range from 0 ("no pain") to 10 ("pain as bad as you can imagine"). BPI also evaluates the degree to which pain has interfered with different areas of participants' lives over the past 24 hours: general activity, walking, work, mood, enjoyment of life, relations with others and sleep. BPI pain interference is scored as the mean of the seven interference items, each of which is scored from zero ("does not interfere") to 10 ("completely interferes"). Finally, BPI also evaluates the amount of relief of pain treatments have provided in the past 24 hours, ranging from 0% ("no relief") to 100% ("complete relief").

SECONDARY OUTCOMES:
To measure the efficacy SP160412 combined with a placebo in the reduction of clinical sign of sunburn | Twice a Day (in the morning and at night) from day 1 to day 5
  To measure the efficacy of SP160412 on Pruritus. 11-point Itch NRS (Appendix I.3. Pruritus Numeric Rating Scale (NRS)); This instrument is presented as a single 11-point numeric scale with scores from 0 to 10, and anchored at 0 representing "No itch" and 10 representing "Worst imaginable itch"
To measure the efficacy of SP160412 for sleep quality | once a day in the morning from day 1 to 5
  To measure the Sleep quality Scale using The 11-point(NRS)) is an unidimensional patient reported outcome (PRO) for quality of sleep. Participants will on a 11-point numeric rating scale ranging from 0 for "Best possible sleep" to 10 for "Worst possible sleep". Used on a daily basis, sleep diaries are reliable and valid instruments for capturing patient reported outcomes. The sleep quality NRS has good psychometric properties.single-item sleep quality NRS was correlated with pain.
To evaluate the number of subject with adverse events | once a day from Days 2 to 8
  To evaluate the Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0, Change From Baseline in Pain Scores on the Visual Analog Scale at evaluate the safety of SP160412 relative to each component alone combined with a placebo based on the incidence of treatment emergent Adverse Events will be recorded in the daily log by the participant and it will be documented at all evaluation visits. Overall incidence of adverse events will be collected for all days of evaluation, from Visit 0 (Day 0) to Visit 6 (Day 8).
Measurement of the evolution of erythema as measured by the Chromameter | at day one and visit at day 5
  To measure the evolution of erythema color by the use of a Chromameter

CONTACTS AND LOCATIONS:
Overall Officials: Gitanjali Petkar, M.D, Principal Investigator — C.I.D.P
Locations (1):
- CIDP, Phoenix, Mauritius

IPD SHARING:
Plan to Share IPD: No